CLINICAL TRIAL: NCT07133360
Title: Cocktail of Vitamin B, Vitamin D and Melatonine VS Ibuprofen in the Surgical Third Molar Extraction. Randomized Clinical Trial
Brief Title: Combination of Mixed Drugs vs Ibuprofen: a Randomized Clinical Trial
Acronym: CoctailRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jesús Torres García Denche, Doctor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-000736-27
Record Dates: First submitted 2025-06-20; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Swelling Lips &Amp; Face; Pain; Trismus
Keywords: Vitamin B; Vitamin D; Melatonine; Ibuprofen; Third Molar
MeSH Terms: conditions — Facies; Pain; Trismus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen 400 (Active Comparator): Three ibuprofen 400 doses
  Interventions: Procedure: Third molar extraction
- Coctail mixed Drugs (Experimental): Vitamin D, Vitamin B and Melatonine at night instead Ibuprofen
  Interventions: Procedure: Third molar extraction

INTERVENTIONS:
Procedure: Third molar extraction — Surgical third molar extraction with conventional medication

SUMMARY:
Combination of vitamins and melatonine compared with the conventional use of ibuprofen after surgical third molar extraction

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, non ibuprofen allergic, presence of impacted lower third molar

Exclusion Criteria:

* Diseases that avoid surgical intervention

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 10 DAYS
  VAS pain scale
Swelling | 7 DAYS
  Face measurement for swelling
Trismus | 7 DAYS
  Opening limitation

SECONDARY OUTCOMES:
Rescue analgesia | 7 DAYS
  Need for more medications
Inflammatory profile | 7 days
  Blood cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided